CLINICAL TRIAL: NCT03511859
Title: Detecting Circulating Tumor Cells (CTCs) and Cell Free DNA (cfDNA) in Peripheral Blood of Breast Cancer (BC) Patients to Develop the Clinical Application for Early Detection and Diagnostics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CellMaxLife (Industry)
Responsible Party: Sponsor
Other Study IDs: CMx-CTC-BC-001
Record Dates: First submitted 2018-04-17; First posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer. Circulating tumor cells. CTCs. Cell free DNA. cfDNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Mammography/ultrasonography confirmed no findings.
- Cancer Group: The biopsy result is breast cancer.

SUMMARY:
Utilization of circulating-tumor-cell (CTC) and cell free DNA (cfDNA) as novel and noninvasive tests for diagnosis confirmation, therapy selection, and cancer surveillance is a rapidly growing area of interest. In the wake of FDA approval of a liquid biopsy test, it is important for clinicians to acknowledge the obvious clinical utility of liquid biopsy for cancer management throughout the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* All subjects need to sign the informed consent form and age is above 20.
* Control group need to have mammogram /ultrasound results category1-3 and confirmed by PI.
* Cancer group subjects with pathology report confirmed to be malignant have not yet done surgery or treatment will be enrolled to the malignant group for analysis

Exclusion Criteria:

* Not willing to sign the informed consent form
* Have been undergone general anesthesia or regional anesthesia in 1 month
* Have been diagnosed with any type of cancer and been treated
* Have been suffering from autoimmune disorder such as SLE and RA
* Have been suffering from chronic infection such as IBD, pancreatitis, COPD or Interstitial pneumonia.
* Have been suffering from acute infection or other infectious diseases in 3 moths such as TB, pneumonia, urinary tract infection, or cellular infection
* Diagnosed with myelodysplastic syndrome or myeloproliferative diseases
* Other condition which may affect the CTC results, when determined by PI can be confirmed by other tests are if necessary

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The objective of this study is to demonstrate that CTC assay counts can distinguish between healthy subjects and malignant breast cancer subjects, including early stage breast cancer subjects. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan